CLINICAL TRIAL: NCT04474509
Title: The ACTyourCHANGE Study Protocol. Promoting a Healthy Lifestyle in Patients With Obesity With Acceptance and Commitment Therapy. A Randomized Controlled Trial
Brief Title: ACTyourCHANGE Study Protocol. Promoting Healthy Lifestyle With ACT for Obesity
Acronym: ACTyourCHANGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03C024
Record Dates: First submitted 2020-07-04; First posted 2020-07-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Health Behavior
Keywords: Acceptance and Commitment Therapy (ACT); Focused-Acceptance and Commitment Therapy (FACT); Obesity; Psychological flexibility; Cognitive Behavioral Therapy (CBT)
MeSH Terms: conditions — Health Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: Three-arm Individually Randomized Group Treatment Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FACT Module Engagement (Experimental): During this module, patients will have the opportunity to increase their motivation to change and encourage the engagement in committed actions, consistent with their life values. Patients are invited to reflect on what is important in their lives, which values make their life worth living, and which actions they could take to live a meaningful life, in accordance with personal values. The use of metaphors and experiential exercises will facilitate the process of exploring personal values, identifying life directions and related behaviors. For example, the 80th Birthday Party metaphor requires participants to imagine there is a party in honor of their birthday and the time comes when people are starting to give speeches and try to answer the question about what they want to hear people at the party say. This exercise help patients in wondering what person they want to be with themselves and others.
  Interventions: Behavioral: FACT Module Engagement
- FACT Module Openness (Experimental): Participants attending this module are guided to recognize and distancing themselves to stressful thoughts, feelings and sensations. They will learn to read suffering as part of human experience, without self-judgment and self-condemnation. Rather, therapist will encourage the patient's assumption of an open and acceptable approach to internal experiences. Throughout the module, therapist will help patients to reflect on their usual, but ineffective efforts to solve personal problems, and encourage the adoption of new responsive strategies based on acceptance and defusion from personal distress.
  An example of metaphor used during the Module is The Passenger on a bus. In this metaphor patient have to imagine to be a driver bus and his every thought is a passenger that gets on and off the bus. This exercise help patients to accept, defuse from, and reduce the power of their thoughts.
  Interventions: Behavioral: FACT Module Openness
- FACT Module Awareness (Experimental): The module comprises meditation exercises and experiences aimed to learn how to act intentionally with awareness about personal thought and sensations without automatically reacting. Participants are supported to recognize their actions and the context where they occur and learn to choose to respond with action consistent with their values and not automatically. Therapist will propose breathing exercises, body scan and others mindfulness experiences. Participants will be encouraged to sitting comfortably, close the eyes, feel themselves in contact with the present moment they are living, paying attention to their breath, noticing the rhythm and any other aspect of the experience of breathing. Then, the therapist guides the participant's attention on the body, noting any part of their body from the head to feet. Then, the sounds around, any noises that could distract their attention on themselves.
  Interventions: Behavioral: FACT Module Awareness

INTERVENTIONS:
Behavioral: FACT Module Engagement — Focused- Acceptance and Commitment Therapy. Third-wave Cognitive Behavioral Therapy (Psychological intervention)
  Arms: FACT Module Engagement
Behavioral: FACT Module Openness — Focused- Acceptance and Commitment Therapy. Third-wave Cognitive Behavioral Therapy (Psychological intervention)
  Arms: FACT Module Openness
Behavioral: FACT Module Awareness — Focused- Acceptance and Commitment Therapy. Third-wave Cognitive Behavioral Therapy (Psychological intervention)
  Arms: FACT Module Awareness

SUMMARY:
Background: as treatment of choice in promoting psychological flexibility, Acceptance and Commitment Therapy (ACT) was found to be effective in several conditions, and among different populations, including weight management in individuals with obesity. However, the mechanism of action of psychological flexibility is less known. The aim of the present study is, within the context of a brief ACT intervention for behavioral change and behavioral maintenance of a healthy lifestyle in a sample of inpatients with obesity, to explore the effect of each subcomponent of the psychological flexibility model on treatment processes and outcomes.

Methods: a randomized controlled trial will be conducted. 90 Italian adult inpatients with obesity attending a rehabilitation program for weight loss will be randomly allocated into three experimental conditions targeting respectively each subcomponent of the psychological flexibility model: group Engage focused on values-oriented behaviors, group Openness focused on acceptance and cognitive defusion, and group Awareness focused on being present and aware of thought, feelings, and behaviors at every moment. Weight, BMI (Kg/m2), the Psychological General Well Being Inventory (PGWBI), the Outcome Questionnaire-45.2 (OQ-45.2), the Depression Anxiety and Stress Scale (DASS-21), the Difficulties in Emotion regulation scale (DERS) the Dutch eating Behaviors Questionnaire (DEBQ), the Brief Values Inventory (BVI), the Committed Action Questionnaire (CAQ), the Italian-Cognitive Fusion Questionnaire (I-CFQ), and the Five Facet Mindfulness Questionnaire (FFMQ) and the Acceptance and Action Questionnaire (AAQ II) will be assessed at the beginning (Time 0), at the end of psychological intervention (Time 1), after 3 (Time 2) and 6 months (Time 3) and 9 months (Time 4) from discharge. During the following month after discharge, outpatients will be monitored in their adherence to a healthy lifestyle, using a wearable device.

To assess the effectiveness of intervention, mixed between-withing 3 (conditions) x 4 (times) repeated measure ANOVAs will be conducted to examine changes from time 0 to time 1, 2, 3 and 4 in means of weight, BMI, and means scores PGWBI, OQ-45.2, DASS; DERS; DEBQ, AAQ-II, BVI, CAQ, I-CFQ, and FFMQ, between three groups Discussion: This study will contribute to clarify the mechanism of action of each subcomponent of the psychological flexibility model and understand its impact on the promotion of a healthy lifestyle.

DETAILED DESCRIPTION:
Obesity is one of the most serious health problems in global public health (Durrer Schutz et al., 2019). Recent estimates pointed out that over the last years obesity reached epidemic proportions, and its prevalence is still rising. In 2016 over 1.9 billion adults in the world were overweight and, of these, more than 650 million were obese (Castelnuovo, Pietrabissa, Manzoni, Cattivelli, Rossi, Novelli, Varallo, 2017).

Defined as an excess of body weight, obesity is a significant risk factor for a plethora of physical, psychological, and social problems, all of which can heavily impact health, quality of life, and global functioning. Obesity is frequently associated with many physical comorbidities, including type II diabetes mellitus, cardiovascular disease, hypertension, kidney failure, and osteoarthritis (Afolabi et al., 2020), psychological problems such as depression, feelings of shame, low self-esteem, stigma (Riva et al., 2006), and eating disorders, as well as social and economic impairment (Kolotkin & Andersen, 2017).

Given the complex nature of the phenomenon, comprehensive multidisciplinary and multi-component lifestyle interventions for the management of obesity in adults are recommended. They include nutrition and dieting, physical activity, and psychological support, aimed at fostering the adoption of a healthy lifestyle through the Cognitive Behavioral Therapy-based interventions considered the gold standard for the treatment of obesity (Giusti et al., 2020).

Even if such programs have been recognized as effective in promoting healthy lifestyle adoption, the maintenance of behavioral change remains challenging. Most obese or overweight people who attend a weight loss rehabilitation program fail to maintain a healthy lifestyle over time. As a consequence, they regain about one-third of the weight lost over the following year after treatment (Castelnuovo & Simpson, 2011; Roberto Cattivelli et al., 2018). This evidence has spurred research to investigate which factors represent barriers to weight loss maintenance and which factors may influence the adoption of healthy lifestyle habits.

Forman and Butryn's conceptual model (Forman & Butryn, 2015) suggest that long-standing adherence to a healthy lifestyle is partially due to some self-regulation skills, such as distress tolerance, values clarity, metacognitive awareness, and behavioral commitment. Such skills were found to play a protective role against the excessive responsiveness to such internal (such as emotions) and external (the availability of tasty food in the modern environment) cues that motivate people to eat palatable food in response to negative internal states, as in case of emotional eating.

Emotional eating refers to eating in response to unpleasant emotional states (Frayn & Knäuper, 2018). Since emotional eating has been associated with elevated consumption of high-calorie and high fat, it doesn't surprise that emotional eating was found to be strongly related to obesity (Konttinen et al., 2010) both in adults and in the younger population (Shapiro et al., 2007;van Strien et al., 2016).

The link between negative emotions and emotional eating has been well-established bot in general (Litwin et al., 2017) and in obese population (Varallo et al., 2021). Many studies suggested that dysfunctional eating habits, such as emotional eating may emerge as a failure of emotion regulation strategies that allow individuals to regulate their own emotions by modulating their responses (Gianini et al., 2013; Stice & Bearman, 2001). As a results, individuals eat as an attempt to regulate their negative internal states.

The treatment of choice to promote self-regulation skills is Acceptance and Commitment Therapy (ACT; Hayes et al., 2006). ACT is one of the recent third-wave Cognitive Behavioral Therapies (CBTs) rised in the last twenty years. It is a transdiagnostic approach aimed at promoting psychological flexibility defined as the ability of "being in contact with the present moment fully as a conscious human being and, basing on what the situation affords, changing or persisting in behavior in the service of chosen values" (Hayes et al., 2006). The promotion of psychological flexibility is based on three subcomponents of the psychological flexibility model: openness, awareness, and engagement. Openness refers to the willingness to develop an open and acceptable attitude toward one's personal internal states such as thoughts, emotions, and bodily sensations; Awareness refers to the ability to act intentionally with awareness about personal thought and sensations, without automatically reacting; Engagement refers to engage oneself in committed behaviors related to personal values, that is chosen life directions (Strosahl et al., 2012).

Over the years, ACT has been successfully applied in various pathological conditions, including obesity management both in adult and young populations (Berman et al., 2016; Levin et al., 2020;Weineland et al., 2012). In an RCT (Cattivelli et al., 2021) comparing a standard CBT-based group psychological intervention with an ACT-based group psychological intervention within an in-hospital multidisciplinary rehabilitation program for weight loss for patients with obesity, it was found that, since there were no significant differences between groups from pre-to post interventions in weight reduction (both groups showed a decrease of weight and BMI from pre to post intervention), only participants in the ACT condition were able to maintain weight lost during the intervention, over the following 6 month after discharge. About the psychological conditions, CBT was greater than ACT in producing improvement in the psychological conditions (subjective well-being, psychological problems, life functioning, risk for self-harm or harm others) from pre-to-post-intervention. On the contrary, at 6 months-follow-up, the effect of the intervention was more extensive in the ACT condition than in CBT. The difference between the two intervention was reasonably attributed to the intrinsic different goals of the therapy: while CBT is focused on the reduction of symptoms (Teixera, Silva, Mata, Palmeira, & Markland., 2012), providing an immediate - but not lasting - relief, ACT fosters psychological flexibility, considered the core mechanism of action of therapy (Hayes et al., 2006).

In the field of health promotion, it was found that psychological flexibility forsters the adoption and the maintenance of beahviors which are driven by personal values and promotes an open, willing and accepting attitude towards internal and external undesirable private events such as thoughts, emotions and bodily sensations. Finally, it improves the ability to be present, in the moment and face events in the context they happen (Butryn et al., 2011).

Even if it has been well-established that psychological flexibility is the core mechanism of action in the ACT-based interventions, less is known about how each subcomponent acts.

To the authors' knowledge, only one study (Villatte et al., 2016) has previously explored the specific effect of two subcomponents of the ACT on treatment processes and outcomes in 15 adult seeking mental health treatment, founding that both the modules - one targeting acceptance and defusion, and one targeting values-based activation - produced improvements in psychiatric symptoms and quality of life, as well as improvements in specific therapeutic processes. However, no study has already assessed the specific effect of every single sub-component of psychological flexibility model, in weight management.

On the basis of these premises, the aim of the current study is to assess - within the context of a brief ACT-based intervention aimed to promote the adoption and maintenance of healthy lifestyle behaviors in a sample of Italian adult individuals with obesity - the specific effect of each subcomponent of the ACT model on the promotion, and most importantly, the maintenance of a healthy lifestyle.

The intervention will be part of a multidisciplinary one-month rehabilitation program for weight loss.

Obesity is one of the most serious health problems in global public health (Durrer Schutz et al., 2019). Recent estimates pointed out that over the last years obesity reached epidemic proportions, and its prevalence is still rising. In 2016 over 1.9 billion adults in the world were overweight and, of these, more than 650 million were obese (Castelnuovo, Pietrabissa, Manzoni, Cattivelli, Rossi, Novelli, Varallo, 2017).

Defined as an excess of body weight, obesity is a significant risk factor for a plethora of physical, psychological, and social problems, all of which can heavily impact health, quality of life, and global functioning. Obesity is frequently associated with many physical comorbidities, including type II diabetes mellitus, cardiovascular disease, hypertension, kidney failure, and osteoarthritis (Afolabi et al., 2020), psychological problems such as depression, feelings of shame, low self-esteem, stigma (Riva et al., 2006), and eating disorders, as well as social and economic impairment (Kolotkin & Andersen, 2017).

Given the complex nature of the phenomenon, comprehensive multidisciplinary and multi-component lifestyle interventions for the management of obesity in adults are recommended. They include nutrition and dieting, physical activity, and psychological support, aimed at fostering the adoption of a healthy lifestyle through the Cognitive Behavioral Therapy-based interventions considered the gold standard for the treatment of obesity (Giusti et al., 2020).

Even if such programs have been recognized as effective in promoting healthy lifestyle adoption, the maintenance of behavioral change remains challenging. Most obese or overweight people who attend a weight loss rehabilitation program fail to maintain a healthy lifestyle over time. As a consequence, they regain about one-third of the weight lost over the following year after treatment (Castelnuovo & Simpson, 2011; Roberto Cattivelli et al., 2018). This evidence has spurred research to investigate which factors represent barriers to weight loss maintenance and which factors may influence the adoption of healthy lifestyle habits.

Forman and Butryn's conceptual model (Forman & Butryn, 2015) suggest that long-standing adherence to a healthy lifestyle is partially due to some self-regulation skills, such as distress tolerance, values clarity, metacognitive awareness, and behavioral commitment. Such skills were found to play a protective role against the excessive responsiveness to such internal (such as emotions) and external (the availability of tasty food in the modern environment) cues that motivate people to eat palatable food in response to negative internal states, as in case of emotional eating.

Emotional eating refers to eating in response to unpleasant emotional states (Frayn & Knäuper, 2018). Since emotional eating has been associated with elevated consumption of high-calorie and high fat, it doesn't surprise that emotional eating was found to be strongly related to obesity (Konttinen et al., 2010) both in adults and in the younger population (Shapiro et al., 2007;van Strien et al., 2016).

The link between negative emotions and emotional eating has been well-established bot in general (Litwin et al., 2017) and in obese population (Varallo et al., 2021). Many studies suggested that dysfunctional eating habits, such as emotional eating may emerge as a failure of emotion regulation strategies that allow individuals to regulate their own emotions by modulating their responses (Gianini et al., 2013; Stice & Bearman, 2001). As a results, individuals eat as an attempt to regulate their negative internal states.

The treatment of choice to promote self-regulation skills is Acceptance and Commitment Therapy (ACT; Hayes et al., 2006). ACT is one of the recent third-wave Cognitive Behavioral Therapies (CBTs) rised in the last twenty years. It is a transdiagnostic approach aimed at promoting psychological flexibility defined as the ability of "being in contact with the present moment fully as a conscious human being and, basing on what the situation affords, changing or persisting in behavior in the service of chosen values" (Hayes et al., 2006). The promotion of psychological flexibility is based on three subcomponents of the psychological flexibility model: openness, awareness, and engagement. Openness refers to the willingness to develop an open and acceptable attitude toward one's personal internal states such as thoughts, emotions, and bodily sensations; Awareness refers to the ability to act intentionally with awareness about personal thought and sensations, without automatically reacting; Engagement refers to engage oneself in committed behaviors related to personal values, that is chosen life directions (Strosahl et al., 2012).

Over the years, ACT has been successfully applied in various pathological conditions, including obesity management both in adult and young populations (Berman et al., 2016; Levin et al., 2020;Weineland et al., 2012). In an RCT (Cattivelli et al., 2021) comparing a standard CBT-based group psychological intervention with an ACT-based group psychological intervention within an in-hospital multidisciplinary rehabilitation program for weight loss for patients with obesity, it was found that, since there were no significant differences between groups from pre-to post interventions in weight reduction (both groups showed a decrease of weight and BMI from pre to post intervention), only participants in the ACT condition were able to maintain weight lost during the intervention, over the following 6 month after discharge. About the psychological conditions, CBT was greater than ACT in producing improvement in the psychological conditions (subjective well-being, psychological problems, life functioning, risk for self-harm or harm others) from pre-to-post-intervention. On the contrary, at 6 months-follow-up, the effect of the intervention was more extensive in the ACT condition than in CBT. The difference between the two intervention was reasonably attributed to the intrinsic different goals of the therapy: while CBT is focused on the reduction of symptoms (Teixera, Silva, Mata, Palmeira, & Markland., 2012), providing an immediate - but not lasting - relief, ACT fosters psychological flexibility, considered the core mechanism of action of therapy (Hayes et al., 2006).

In the field of health promotion, it was found that psychological flexibility forsters the adoption and the maintenance of beahviors which are driven by personal values and promotes an open, willing and accepting attitude towards internal and external undesirable private events such as thoughts, emotions and bodily sensations. Finally, it improves the ability to be present, in the moment and face events in the context they happen (Butryn et al., 2011).

Even if it has been well-established that psychological flexibility is the core mechanism of action in the ACT-based interventions, less is known about how each subcomponent acts.

To the authors' knowledge, only one study (Villatte et al., 2016) has previously explored the specific effect of two subcomponents of the ACT on treatment processes and outcomes in 15 adult seeking mental health treatment, founding that both the modules - one targeting acceptance and defusion, and one targeting values-based activation - produced improvements in psychiatric symptoms and quality of life, as well as improvements in specific therapeutic processes. However, no study has already assessed the specific effect of every single sub-component of psychological flexibility model, in weight management.

On the basis of these premises, the aim of the current study is to assess - within the context of a brief ACT-based intervention aimed to promote the adoption and maintenance of healthy lifestyle behaviors in a sample of Italian adult individuals with obesity - the specific effect of each subcomponent of the ACT model on the promotion, and most importantly, the maintenance of a healthy lifestyle.

The intervention will be part of a multidisciplinary one-month rehabilitation program for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30;
* Written and informed consent to participate; 4) being technology friendly to use wearable devices.

Exclusion Criteria:

* other psychiatric disturbances (diagnosed according to DSM 5 criteria);
* other medical conditions not related to obesity that could compromise participation at the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Weight | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The primary outcome of the study is weight loss maintenance. Weight, and height will be assessed to calculate Body Mass Index (BMI= kg/m2). Weight loss maintenance will be assessed considering the difference between initial weight and weight recorded at follow-up. Success in long term weight loss maintenance is achieved if individual loss at list 10% of initial weight, and maintains weight lost for one year (R. R Wing & Hill, 2001)
Change in Psychological Well-Being | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The second outcome measure is psychological well-being. The Psychological General Well-Being Inventory (PGWBI; (Dupuy, 1984) Italian validation of Grossi and colleagues (Grossi et al., 2006) consist of 22 self-administered items rated on a 6-point Likert scale, relative to six subscales that offer a measure of the level of subjective psychological well-being. Subscales are anxiety, depression, positive well-being, self-control, general health, and vitality with a range of Alpha's scores from 0.61 to 0.85 for each subscale.
Change in Psychological Treatment | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The third outcome measure is the outcome of psychological treatment. The Outcome Questionnaire-45.2 (Lambert, Gregersen, & Burlingame, 2004) Italian version by Chiappelli, Coco, Gullo, Bensi, e Prestano (2008) as a measure for the assessment of psychological treatment is a self-report questionnaire composed by 45 items. Subscales are symptoms distress, interpersonal relations and social role functioning. Total Alpha score is excellent (.90 for clinical sample; .92 for non-clinical sample)

SECONDARY OUTCOMES:
Values | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The Brief Values Inventory (McCracken & Yang, 2006) Italian validation of Baroni, McCracken, Matera, Nerini, & Stefanile ( 2019). It is composed by 12 items aimed to assess the success in living according to personal values. The internal consistency of the Success subscale is .70 in the Italian validation study.
Committed Actions | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The Committed Action Questionnaire (McCracken, 2013) Italian adaptation of Baroni, Matera, Nerini, & Stefanile ( 2017) is 8-items self-report questionnaire rated on 7-point Likert scale, used to assess positive and negative aspects of the ability to engage themselves into committed actions driven by values. The internal consistency of the measure tested on a normative sample was good (α= .80).
Cognitive Fusion | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The Italian-Cognitive Fusion Questionnaire (Gillanders et al., 2014) Italian version by Oppo and colleagues (2019) is 7-items questionnaire administered for the assessment of cognitive fusion. The internal consistency of the Italian version is excellent (α= .82).
Acceptance | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The subscale "Nonjudge" of the Five Facet Mindfulness Questionnaire, described below, is used as a measure of Acceptance. The internal consistency of the subscale is .86
Awareness | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The Five Facet Mindfulness Questionnaire (FFMQ; (Baer, Smith, Hopkins, Krietemeyer, & Toney, 2006). The Italian version (Boffito et al., 2009) is 39-item-self-report questionnaire used as a measure of Mindfulness. It is composed by five subscales: observe, describe, act with awareness, non-react, nonjudge. The internal consistency of total scale is good (α .86).
Psychological inflexibility and experiential avoidance | Baseline, after 4 weeks (Time 1), after 6 months (Time 2), after 1 year (Time 3)
  The Acceptance and Action Questionnaire (AAQ II: (Bond et al., 2011). The Italian version (Pennato, Berrocal, Bernini, & Rivas, 2013) is the most widely used self-reported questionnaire that measures psychological inflexibility and experiential avoidance. It is composed by 10 items, rated on 7-point Likert scale, the Internal consistency is good (α .83) and test-retest reliability is moderate (.61)

CONTACTS AND LOCATIONS:
Locations (1):
- San Giuseppe Hospital, Istituto Auxologico Italiano IRCSS, Verbania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fairburn CG, Rothwell ER. Apps and eating disorders: A systematic clinical appraisal. Int J Eat Disord. 2015 Nov;48(7):1038-46. doi: 10.1002/eat.22398. Epub 2015 Feb 27. PMID 25728705
- [Background] Cattivelli R, Pietrabissa G, Ceccarini M, Spatola CA, Villa V, Caretti A, Gatti A, Manzoni GM, Castelnuovo G. ACTonFOOD: opportunities of ACT to address food addiction. Front Psychol. 2015 Apr 9;6:396. doi: 10.3389/fpsyg.2015.00396. eCollection 2015. No abstract available. PMID 25914662
- [Result] Villatte JL, Vilardaga R, Villatte M, Plumb Vilardaga JC, Atkins DC, Hayes SC. Acceptance and Commitment Therapy modules: Differential impact on treatment processes and outcomes. Behav Res Ther. 2016 Feb;77:52-61. doi: 10.1016/j.brat.2015.12.001. Epub 2015 Dec 10. PMID 26716932
- [Result] Forman EM, Butryn ML, Manasse SM, Crosby RD, Goldstein SP, Wyckoff EP, Thomas JG. Acceptance-based versus standard behavioral treatment for obesity: Results from the mind your health randomized controlled trial. Obesity (Silver Spring). 2016 Oct;24(10):2050-6. doi: 10.1002/oby.21601. PMID 27670400
- [Derived] Guerrini Usubini A, Cattivelli R, Giusti EM, Riboni FV, Varallo G, Pietrabissa G, Manzoni GM, Consoli S, Bastoni I, Granese V, Volpi C, Villa V, Caretti A, Bottacchi M, Castelnuovo G, Molinari E. The ACTyourCHANGE study protocol: promoting a healthy lifestyle in patients with obesity with Acceptance and Commitment Therapy-a randomized controlled trial. Trials. 2021 Apr 20;22(1):290. doi: 10.1186/s13063-021-05191-y. PMID 33879183